CLINICAL TRIAL: NCT04064515
Title: Identification of Circulating Tumor Cells in Patients With HPV 16 or 18 Associated Cervical Cancer
Brief Title: CTCs in Cervix Cancer
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 19-00495
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Cervical Cancer; HPV
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA will be used to test CTCs identified for the presence of the HPV 16 / 18 E6 protein, confirming a cervical cancer origin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cervical Cancer: Participants with advanced or recurrent cervical cancer will provide 15 mL of whole blood. Participants will then be followed prospectively for three years to document oncologic outcome.
  Interventions: Diagnostic Test: Blood Assayed for CTCs
- Control: Participants without a history of cervical cancer or high grade pre-cancer of the cervix
  Interventions: Diagnostic Test: Blood Assayed for CTCs

INTERVENTIONS:
Diagnostic Test: Blood Assayed for CTCs — All study participants will have 15 mL of blood drawn for the purpose of the study.

SUMMARY:
This study is a validation study to confirm the ability of Telomescan OBP-401 to identify CTCs in patients with HPV 16 / 18 associated cervical cancer. CTCs identified will be tested for the presence of the HPV 16 / 18 E6 protein, confirming a cervical cancer origin.

ELIGIBILITY:
Inclusion Criteria:

* Able to safely provide 15 ml of blood
* Able to provide informed consent
* Pathologically confirmed invasive cervical cancer
* Proof of serotype HPV 16 or HPV 18 positive within 3 years of the study
* Patients with stages IIA2 to IVB OR recurrent cervical cancer
* For patients with newly diagnosed cervical cancer, they must be enrolled (blood drawn) prior to initiating anti-cancer therapy
* For patients with recurrent cervical cancer, they must be enrolled (blood drawn) prior to initiating a new anti-cancer therapy for progression of disease (based on RECIST 1.1 criteria). Patients who have progressed and are moving to best supportive care are eligible.
* If patients meet criteria 5.1A 5 above, the following criteria must be met:
* At least 21 days have elapsed following treatment with cytotoxic chemotherapy
* At least 14 days have elapsed following treatment with biologic therapy
* At least 14 days have elapsed following radiation therapy

Exclusion Criteria:

* History of any cancer other than cervix cancer within the past five years.
* History of any known germ-line pathogenic mutation (ie BRCA 1 / 2 or Lynch syndrome, but genetic testing is not required)
* Current use of systemic corticosteroids at doses exceeding 10 mg per day of prednisone or its equivalent.
* Active infection including hepatitis B, hepatitis C, HIV.
* Any patient unable to comply with the study criteria.
* Patients taking any anti-inflammatory agents (aspirin, NSAIDs, steroids), within 24 hrs prior to blood draw.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman age 18 or older, with pathologically confirmed invasive cervical cancer
Study Population: Two groups will be recruited: the case group will consist of 16 participants with advanced or recurrent cervical cancer; the control arm will consist of 16 participants without a history of cervical cancer or high grade pre-cancer of the cervix.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Effectiveness of OBP-401 to identify CTCs in patients with active HPV 16 / 18 associated cervical cancer compared to non-cancer controls (patients without CIN 2 - 3 or cancer). | 3 Years

SECONDARY OUTCOMES:
Presence of HPV 16 or 18 genome in the samples with a positive CTC result, in order to confirm a cervical cancer origin. | 3 Years
Recurrence rates in patients stratified by CTC identification | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Boyd, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States